CLINICAL TRIAL: NCT03449082
Title: Treatment of Intractable Common Extensor Tendon Injury Using Allogeneic Adipose-derived Mesenchymal Stem Cells (Allo-ASC): a Phase II Randomized Controlled Trial
Brief Title: Treatment of Intractable Common Extensor Tendon Injury Using Mesenchymal Stem Cells (Allo-ASC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUH-RM-SGChung-ASC-02
Record Dates: First submitted 2018-01-30; First posted 2018-02-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Lateral Epicondylitis
Keywords: adipose derived mesenchymal stem cell; allogeneic stem cell
MeSH Terms: conditions — Tennis Elbow | interventions — Fibrin Tissue Adhesive; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High concentration of Allo-ASC group (Experimental): High concentration of Allo-ASC 0.5cc (Total: 10 million cells) & Fibrin glue 0.5cc by ultrasonographic guided intra-tendon injection
  Interventions: Biological: High concentration of Allo-ASC; Drug: Fibrin glue
- Low concentration of Allo-ASC group (Experimental): Low concentration of Allo-ASC 0.5cc (Total: 1 million cells) & Fibrin glue 0.5cc by ultrasonographic guided intra-tendon injection
  Interventions: Biological: Low concentration of Allo-ASC; Drug: Fibrin glue
- Placebo Comparator (Fibrin) group (Placebo Comparator): Normal saline 0.5cc & Fibrin glue 0.5cc by ultrasonographic guided intra-tendon injection
  Interventions: Drug: Fibrin glue; Drug: Normal saline

INTERVENTIONS:
Biological: High concentration of Allo-ASC — 10 million cells of Allo-ASC 0.5cc
  Arms: High concentration of Allo-ASC group
Biological: Low concentration of Allo-ASC — 1 million cells of Allo-ASC 0.5cc
  Arms: Low concentration of Allo-ASC group
Drug: Fibrin glue — Fibrin glue 0.5cc
  Other Names: Fibrin sealant
Drug: Normal saline — Normal saline 0.5cc
  Other Names: 0.9% Sodium Chloride Solution
  Arms: Placebo Comparator (Fibrin) group

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intra-tendon injection of allogeneic adipose-derived mesenchymal stem cells (Allo-ASC) in intractable common extensor tendinosis patients in comparison with a control treatment.

DETAILED DESCRIPTION:
A phase II randomized placebo controlled trial will be done with following 3 groups. Each group will have 10 participants, so, the total patients will be 30 people.

1. High concentration of Allo-ASC group: stem cell 0.5cc (Total: 10 million cells) + Fibrin glue 0.5cc
2. Low concentration of Allo-ASC group: stem cell 0.5cc (Total: 1 million cells) + Fibrin glue 0.5cc
3. Placebo Comparator (Fibrin) group: Normal saline 0.5cc + Fibrin glue 0.5cc The investigators will compare the efficacy difference with visual analogue scale (VAS) during activity (primary outcome), VAS at rest, Mayo elbow performance index (MEPI), grip strength, ultrasonographic assessment at baseline, 6 weeks, 12 weeks, 6 months, 12 months and 24 months after injection. Shear wave elastography (SWE) and magnetic resonance image (MRI) will be done at baseline, 12 weeks, 12 months and 24 months after injection

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as lateral epicondylosis (tennis elbow)
* symptom duration is over 12 months
* pain visual analogue scale (VAS) during activity ≥ 5
* recurrent pain in spite of conservative treatment such as physical therapy, medication, steroid injection
* common extensor tendon injury can be observed under ultrasound (hypoechoic lesion) and MRI (hyperintensity or discontinuity)
* patient that can understand the clinical trials

Exclusion Criteria:

* patient that underwent other injection such as steroid injection or prolotherapy within 6 weeks
* patients with following conditions (such as arthritis related to the target lesion, synovitis related to the target lesion, paralysis related to the target lesion, entrapment of related nerve to the target lesion, radiculopathy related to the target lesion, infectious disease, generalized pain syndrome, rheumatoid arthritis, impaired sensibility, dementia, history of allergic or hypersensitive reaction to bovine-derived proteins or Fibrin Glue, contraindication to MRI)
* patient that enrolled other clinical trials within 30 days
* current pregnancy or breast-feeding, planning for pregnancy
* history of drug/alcohol addiction, habitual smoker
* operation history of affected elbow
* previous clinical trial involving stem cell administration
* other severe medical illness or bleeding tendency
* size of intramural calcification over 2.0 mm under ultrasound evaluation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Change of pain visual analogue scale (VAS) during activity | baseline and 12 weeks
  Self reported pain intensity during activity will be evaluated by visual analogue scale (0 = no pain, 10 = pain as bad as can be).

SECONDARY OUTCOMES:
Change of pain visual analogue scale (VAS) during activity | baseline, 6 weeks, 12 weeks, 6 months, 12 months and 24 months
  Self reported pain intensity during activity will be evaluated by visual analogue scale (0 = no pain, 10 = pain as bad as can be).
Change of pain visual analogue scale (VAS) at rest | baseline, 6 weeks, 12 weeks, 6 months, 12 months and 24 months
  Self reported pain intensity at rest will be evaluated by visual analogue scale (0 = no pain, 10 = pain as bad as can be).
Change of Mayo elbow performance index (MEPI) | baseline, 6 weeks, 12 weeks, 6 months, 12 months and 24 months
  The MEPI measures pain, motion, stability, and daily functions. (0 = worst, 100 = best)
Ultrasonographic assessment | baseline, 6 weeks, 12 weeks, 6 months, 12 months and 24 months
  Ultrasonographic findings will be analyzed using a 5-point Likert scale (1: more aggravated, 2: aggravated, 3: same, 4: improved, 5: more improved). Sonographic images will be compared with baseline images by experienced ultrasound examiners being blind to the treatment group and the time points of image achievement.
Shear wave elastography | baseline, 12 weeks and 24 months
  Young modulus and shear wave speed will be obtained
Magnetic resonance image (MRI) assessment | baseline, 12 weeks and 24 months
  MRI findings will be analyzed using a 5-point Likert scale (1: more aggravated, 2: aggravated, 3: same, 4: improved, 5: more improved). MR images will be compared with baseline images by experienced ultrasound examiners being blind to the treatment group and the time points of image achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gun Chung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SY, Kim W, Lim C, Chung SG. Treatment of Lateral Epicondylosis by Using Allogeneic Adipose-Derived Mesenchymal Stem Cells: A Pilot Study. Stem Cells. 2015 Oct;33(10):2995-3005. doi: 10.1002/stem.2110. Epub 2015 Aug 6. PMID 26202898
- [Background] Lee SY, Kwon B, Lee K, Son YH, Chung SG. Therapeutic Mechanisms of Human Adipose-Derived Mesenchymal Stem Cells in a Rat Tendon Injury Model. Am J Sports Med. 2017 May;45(6):1429-1439. doi: 10.1177/0363546517689874. Epub 2017 Mar 14. PMID 28291954
- [Background] Pascual-Garrido C, Rolon A, Makino A. Treatment of chronic patellar tendinopathy with autologous bone marrow stem cells: a 5-year-followup. Stem Cells Int. 2012;2012:953510. doi: 10.1155/2012/953510. Epub 2011 Dec 18. PMID 22220180
- [Background] Ellera Gomes JL, da Silva RC, Silla LM, Abreu MR, Pellanda R. Conventional rotator cuff repair complemented by the aid of mononuclear autologous stem cells. Knee Surg Sports Traumatol Arthrosc. 2012 Feb;20(2):373-7. doi: 10.1007/s00167-011-1607-9. Epub 2011 Jul 20. PMID 21773831
- [Background] Hernigou P, Flouzat Lachaniette CH, Delambre J, Zilber S, Duffiet P, Chevallier N, Rouard H. Biologic augmentation of rotator cuff repair with mesenchymal stem cells during arthroscopy improves healing and prevents further tears: a case-controlled study. Int Orthop. 2014 Sep;38(9):1811-8. doi: 10.1007/s00264-014-2391-1. Epub 2014 Jun 7. PMID 24913770
- [Background] Zhang X, Lin YC, Rui YF, Xu HL, Chen H, Wang C, Teng GJ. Therapeutic Roles of Tendon Stem/Progenitor Cells in Tendinopathy. Stem Cells Int. 2016;2016:4076578. doi: 10.1155/2016/4076578. Epub 2016 Apr 19. PMID 27195010
- [Background] Clarke AW, Alyas F, Morris T, Robertson CJ, Bell J, Connell DA. Skin-derived tenocyte-like cells for the treatment of patellar tendinopathy. Am J Sports Med. 2011 Mar;39(3):614-23. doi: 10.1177/0363546510387095. Epub 2010 Dec 7. PMID 21139155
- [Background] Leong DJ, Sun HB. Mesenchymal stem cells in tendon repair and regeneration: basic understanding and translational challenges. Ann N Y Acad Sci. 2016 Nov;1383(1):88-96. doi: 10.1111/nyas.13262. Epub 2016 Oct 5. PMID 27706825
- [Background] Muller SA, Todorov A, Heisterbach PE, Martin I, Majewski M. Tendon healing: an overview of physiology, biology, and pathology of tendon healing and systematic review of state of the art in tendon bioengineering. Knee Surg Sports Traumatol Arthrosc. 2015 Jul;23(7):2097-105. doi: 10.1007/s00167-013-2680-z. Epub 2013 Sep 21. PMID 24057354
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Maffulli N, Longo UG, Denaro V. Novel approaches for the management of tendinopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2604-13. doi: 10.2106/JBJS.I.01744. PMID 21048180
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Tobita M, Orbay H, Mizuno H. Adipose-derived stem cells: current findings and future perspectives. Discov Med. 2011 Feb;11(57):160-70. PMID 21356171
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Chong AK, Ang AD, Goh JC, Hui JH, Lim AY, Lee EH, Lim BH. Bone marrow-derived mesenchymal stem cells influence early tendon-healing in a rabbit achilles tendon model. J Bone Joint Surg Am. 2007 Jan;89(1):74-81. doi: 10.2106/JBJS.E.01396. PMID 17200313
- [Background] Nixon AJ, Dahlgren LA, Haupt JL, Yeager AE, Ward DL. Effect of adipose-derived nucleated cell fractions on tendon repair in horses with collagenase-induced tendinitis. Am J Vet Res. 2008 Jul;69(7):928-37. doi: 10.2460/ajvr.69.7.928. PMID 18593247
- [Background] Guadalajara H, Herreros D, De-La-Quintana P, Trebol J, Garcia-Arranz M, Garcia-Olmo D. Long-term follow-up of patients undergoing adipose-derived adult stem cell administration to treat complex perianal fistulas. Int J Colorectal Dis. 2012 May;27(5):595-600. doi: 10.1007/s00384-011-1350-1. Epub 2011 Nov 9. PMID 22065114
- [Background] Guest DJ, Smith MR, Allen WR. Monitoring the fate of autologous and allogeneic mesenchymal progenitor cells injected into the superficial digital flexor tendon of horses: preliminary study. Equine Vet J. 2008 Mar;40(2):178-81. doi: 10.2746/042516408X276942. PMID 18267891
- [Background] Hohendorff B, Siepen W, Spiering L, Staub L, Schmuck T, Boss A. Long-term results after operatively treated Achilles tendon rupture: fibrin glue versus suture. J Foot Ankle Surg. 2008 Sep-Oct;47(5):392-9. doi: 10.1053/j.jfas.2008.05.006. Epub 2008 Jul 14. PMID 18725118
- [Background] Smidt N, van der Windt DA, Assendelft WJ, Deville WL, Korthals-de Bos IB, Bouter LM. Corticosteroid injections, physiotherapy, or a wait-and-see policy for lateral epicondylitis: a randomised controlled trial. Lancet. 2002 Feb 23;359(9307):657-62. doi: 10.1016/S0140-6736(02)07811-X. PMID 11879861
- [Background] Jindal N, Gaury Y, Banshiwal RC, Lamoria R, Bachhal V. Comparison of short term results of single injection of autologous blood and steroid injection in tennis elbow: a prospective study. J Orthop Surg Res. 2013 Apr 27;8:10. doi: 10.1186/1749-799X-8-10. PMID 23621906
- [Background] Jacobson JA, Chiavaras MM, Lawton JM, Downie B, Yablon CM, Lawton J. Radial collateral ligament of the elbow: sonographic characterization with cadaveric dissection correlation and magnetic resonance arthrography. J Ultrasound Med. 2014 Jun;33(6):1041-8. doi: 10.7863/ultra.33.6.1041. PMID 24866611
- [Background] Scutt N, Rolf CG, Scutt A. Glucocorticoids inhibit tenocyte proliferation and Tendon progenitor cell recruitment. J Orthop Res. 2006 Feb;24(2):173-82. doi: 10.1002/jor.20030. PMID 16435354
- [Background] Dirrichs T, Quack V, Gatz M, Tingart M, Rath B, Betsch M, Kuhl CK, Schrading S. Shear Wave Elastography (SWE) for Monitoring of Treatment of Tendinopathies: A Double-blinded, Longitudinal Clinical Study. Acad Radiol. 2018 Mar;25(3):265-272. doi: 10.1016/j.acra.2017.09.011. Epub 2017 Nov 16. PMID 29153963
- [Background] Domenichini R, Pialat JB, Podda A, Aubry S. Ultrasound elastography in tendon pathology: state of the art. Skeletal Radiol. 2017 Dec;46(12):1643-1655. doi: 10.1007/s00256-017-2726-2. Epub 2017 Aug 1. PMID 28765991